CLINICAL TRIAL: NCT01516593
Title: Phase II Study on Safety and Activity of a Short Term Intensified Chemo-immunotherapy Combination in HIV-positive Patients Affected by Burkitt Lymphoma
Brief Title: Short Term Intensified Chemo-immunotherapy in HIV-positive Patients With Burkitt Lymphoma
Acronym: CARMEN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andres J. M. Ferreri (Other)
Responsible Party: Sponsor-Investigator, Andres J. M. Ferreri, MD, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARMEN
Record Dates: First submitted 2012-01-06; First posted 2012-01-25 (Estimated); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: HIV; Burkitt's Lymphoma
Keywords: HIV; Burkitt's lymphoma; intensive; short term; immuno-chemotherapy; HIV-positive patients with Burkitt's lymphoma
MeSH Terms: conditions — Burkitt Lymphoma | interventions — Cytarabine; Transplantation Conditioning; Transplantation, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intensive short term immuno-chemotherapy (Experimental): Experimental treatment consists of an induction phase followed by a consolidation or intensified phase according to tumor response.
  Interventions: Drug: Induction Phase; Drug: Consolidation Phase (on day +50); Drug: Intensification phase; Drug: BEAM conditioning; Radiation: Consolidation radiotherapy

INTERVENTIONS:
Drug: Induction Phase — * dd -2 to 1: Methylprednisolone
  * dd 0-1, Cyclophosphamide, associated on day 0 with Vincristine
  * dd 2, Rituximab
  * dd 7, Methotrexate
  * dd 14, Rituximab
  * dd 15, Etoposide
  * dd 21, Methotrexate
  * dd 29, Rituximab and Doxorubicin
  * dd 36, Rituximab and VCR
  At the end of this induction phase, subsequent treatment will be performed according to the objective response:
  1. pts in CR: consolidation phase followed by bulky site irradiation
  2. pts in PR: consolidation phase followed by BEAM conditioning regimen supported by ASCT and bulky irradiation
  3. pts with SD after induction or PD during or after induction: intensification phase followed by BEAM conditioning regimen supported by ASCT and bulky irradiation
  Other Names: Short-term intensive sequential chemoimmunotherapy
Drug: Consolidation Phase (on day +50) — * dd 1-2: cytarabine twice a day
  * dd 3 and 11: rituximab
  * dd 11-13: leukapheresis for PBPC collection.
  Other Names: high-dose cytarabine; consolidation phase
Drug: Intensification phase — 1. One or two courses of R-IVAC or R-ICE chemoimmunotherapy regimen, every three weeks as debulking.
  2. CTX (dd 1) associated with rituximab on dd 3 and 10, followed by PBPC collection (dd 11-13);
  3. AraC every 12 hours for four days (dd -5 to -2) supported by reinfusion of CD34+ cells (dd 0), rituximab infusion (dd -1 and +11) and second in-vivo purged PBPC collection (if needed).
  Other Names: unresponsive patients, refractory disease
Drug: BEAM conditioning — BCNU on dd 1; VP-16 every 12 hours on dd 2-5 and araC every 12 hours on dd 2-5; melphalan on dd 6, followed by the reinfusion of CD34+ cells
  Other Names: Conditioning regimen, autologous transplantation
Radiation: Consolidation radiotherapy — At the end of the whole program, patients will be evaluated for involved-field irradiation with 6-10 MeV photons and a dose of 36 Gy (2 Gy/d, five fractions a week). Three subgroups of patients will be considered for radiotherapy
  Other Names: bulky irradiation; residual lesion

SUMMARY:
This is a multicenter,open-label trial to evaluate activity and safety of the investigational intensive in HIV+ patients with Burkitt's lymphoma.

Experimental treatment consists of an induction phase followed by a consolidation or intensified phase according to tumor response.

Until recently, the immuno-compromised state of patients with concomitant HIV/AIDS and BL was thought to limit the ability to administer intensive chemotherapeutic regimens due to infection rate. However, the advent of highly active antiretroviral therapy (HAART) and evidence in diffuse large B-cell lymphomas that HIV-positive patients can tolerate standard chemotherapeutic regimens with improved outcomes have led investigators to treat HIV-positive patients with the same intensive chemotherapy regimens used to treat immuno-competent patients. Data suggest that these current approaches, along with supportive care, may result in improved patient outcomes, similar to those in the immuno-competent patient population.

DETAILED DESCRIPTION:
The activity of feasibility of the proposed program will be assessed in HIV+ patients with Burkitt lymphoma with the aim to improve tolerability, minimize source consuming and supporting treatment and redu ce late sequels. Available combinations in this setting are really source demanding and toxic combinations showing high rates of septic complication and a treatment-related mortality of near 20%.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of Burkitt's lymphoma (WHO 2008)
* HIV sero-positivity
* Age ≥18 and ≤60 years
* ECOG-PS ≤3

Exclusion Criteria:

* CNS parenchymal involvement
* Absolute neutrophil count <1.000 cells/μL and platelets count <75 × 109/L (Burkitt unrelated)
* Creatinine >1,5N (Burkitt unrelated)
* SGOT and/or SGTP >2,5N (Burkitt unrelated)
* Bilirubin >2N (Burkitt unrelated)
* Severe psychiatric illness or any other clinical, social or psychological condition that could interfere with patient's adherence and compliance
* Significant cardiac disease or acute myocardial infarction in the last 12 months
* Severe active infection (except for HBV and/or HCV co-infection)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2011-11; Primary Completion 2013-04 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
evaluation of activity of the induction phase in terms of complete remission rate | at the end of the induction phase of the investigational intensive chemotherapy, an expected average of 45 days
  Objective lymphoma response achieved after the induction phase of the experimental treatment.

SECONDARY OUTCOMES:
Feasibility and tolerability of the investigational intensive chemotherapy in terms of grade ≥4 adverse events | participants will be followed for the duration of the whole experimental program, an expected average of 100 days
  Assessment of incidence of grade 4 AE during experimental treatment (induction, consolidation and intensification phases as well as conditioning and autologous stem cell transplantation (if indicated)
Feasibility and tolerability of the consolidation phase followed by BEAM conditioning and autologous stem cell transplantation in terms of prevalence of grade ≥4 adverse events | participants will be followed for the duration of the whole experimental program, an expected average of 100 days
Feasibility and tolerability of intensification phase in terms of prevalence of grade ≥4 adverse events | participants will be followed for the duration of the whole experimental program, an expected average of 100 days
  Participants who will not achieve a complete or partial response after induction and consolidation phases will be referred to intensification phase, which will be followed by BEAM + ASCT. These patients will be assess for tolerabbility and AE during these therapeutic phases.
Activity of the whole investigational program in terms of complete remission rate | at the end of the whole program, an expected average of 100 days
  Participants will be assessed by conventional exams to define complete remission rate after the whole experiemntal program; that is after consolidation phase for patients who achieved complete remission after induction phase, after BEAM + ASCt for patients who achieved partial response after induction phase, and after intensification phase for patients who did not achieve an objective response after induction phase.

CONTACTS AND LOCATIONS:
Overall Officials: Andrés JM Ferreri, MD, Study Chair — San Raffaele Scientific Institute, Milano, Italy
Locations (8):
- Italy (8):
  - Oncologia Medica A - Centro di Riferimento Oncologico, Aviano (PN)
  - Ematologia - A.O. Spedali Civili, Brescia
  - Dip. Oncoematologia - Fondazione Centro San Raffaele del Monte Tabor, Milan
  - S.C. Oncologia Medica - Ospedale San Paolo, Milan
  - S.C. Oncologia Medica 3 - IRCCS Istituto Nazionale Tumori (INT), Milan
  - U.O.C. Immunodeficienze virali - I.N.M.I. L. Spallanzani, Roma
  - S.C. Oncoematologia - A.O. Santa Maria, Terni
  - U.O. Ematologia 2 - Ospedale San Giovanni Battista, Torino